CLINICAL TRIAL: NCT07248124
Title: Pilot Study, Aimed at Describing in Myography, the Collapse of the Muscular Response Visualized in the Scratch Collapse Test, in Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SC-My; 2025-A01019-40 (Other: ID-RCB)
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Carpal Tunnel Syndrome (CTS)
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with unilateral carpal tunnel syndrome (Experimental): Patient with clinical unilateral carpal tunnel syndrome diagnosed by history, clinical examination and electromyography,
  Interventions: Procedure: electromyograph; Diagnostic Test: Scratch Collapse Test

INTERVENTIONS:
Procedure: electromyograph — This examination uses electrodes placed along the path of the median nerve to measure the transmission of nerve impulses (conduction studies). It is performed on both hands to compare the results.
Diagnostic Test: Scratch Collapse Test — The Scratch Collapse Test (SCT) is a neurocutaneous reflex used to detect peripheral nerve compression in nerve canal syndromes. It involves first performing a sensory stimulus on the skin at the suspected nerve compression site, then bilaterally testing the strength of a specific muscle in the patient. Compression is then manifested by a transient loss of strength in the muscle on the affected side, while it is preserved on the stimulated side.

SUMMARY:
The Scratch Collapse Test (SCT) is a neurocutaneous reflex used to detect peripheral nerve compression in nerve tunnel syndromes. It first involves applying a sensory stimulus to the skin over the suspected nerve compression point, then bilaterally testing the strength of a specific muscle in the patient. Compression is then manifested by a transient loss of strength in the muscle on the affected side, while it is preserved on the healthy side. This loss of strength is transient and disappears after a few seconds. This test can be performed during a patient's clinical examination, with the physician assessing strength or, conversely, muscle collapse. However, while several articles have described the relevance of this test, as well as its sensitivity and specificity, no study has specifically investigated and measured this observed loss of eccentric muscle tone and its unilateral and transient nature, even though the phenomenon of CSP (cutaneous silent period) has been described.

We therefore propose to analyze the myographic tracing obtained in patients diagnosed with unilateral carpal tunnel syndrome. A transient loss of muscle tone is expected by selective needle myography on the pathological side after cutaneous sensory stimulation of the wrist, while cutaneous sensory stimulation on the healthy side does not alter the tracings obtained by myography.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with clinical unilateral carpal tunnel syndrome diagnosed by history, clinical examination and electromyography,
* Patient who has been informed and has given their free, informed, and written consent,
* Patient affiliated with or beneficiary of a social security scheme.

Exclusion Criteria:

* Other associated canal syndrome on either side (ulnar, defilement, lacertus),

  * Rotator cuff pathology, insufficiency or rupture of the infraspinatus,
  * Associated cervical pathology,
  * Neuropathy, central or peripheral neurological disease,
  * Diabetic patient,
  * Patient with cognitive impairments that prevent the understanding of the study information,
  * Refusal to participate in the study,
  * Pregnant, parturient, or breastfeeding woman,
  * Patient under legal protection,
  * Patient not receiving health protection,
  * Protected patient: adult under guardianship, curatorship, or other legal protection, deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Evolution of the myographic tracings | one day
  Evolution of the myographic tracings (of the infraspinatus muscle) of the pathological arm immediately after ipsilateral stimuli compared to the basic tracings (before stimuli) of the pathological arm and evolution of the myographic tracings of the pathological arm 20 seconds after ipsilateral stimuli compared to the basic tracings (before stimuli) of the pathological arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de l'Ormeau, Tarbes, France